CLINICAL TRIAL: NCT01878578
Title: The Effect of BIA 2-093 on the Steady-state Pharmacokinetic Profile of Phenytoin in Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: prematurely terminated due to impossibility of recruiting the planned number of patients by the study centre.
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIA-2093-106
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Epilepsy
Keywords: Anticonvulsant, BIA 2-093
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Phenytoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eslicarbazepine acetate (Experimental): ESL 600 mg tablets
  Interventions: Drug: Eslicarbazepine acetate
- phenytoin (Active Comparator): Hidantina® 100 mg tablets
  Interventions: Drug: phenytoin
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eslicarbazepine acetate — Tablets containing ESL 600 mg
  Other Names: BIA 2-093
  Arms: Eslicarbazepine acetate
Drug: phenytoin — Hidantina® tablets containing 100 mg of phenytoin
  Other Names: Hidantina® 100 mg tablets
  Arms: phenytoin
Drug: Placebo — Tablets containing matching placebo
  Other Names: Placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is determine the interaction of eslicarbazepine acetate (ESL, BIA 2-093) on the steadystate pharmacokinetics of phenytoin in patients and to evaluate the tolerability and safety of ESL administered concomitantly with phenytoin in patients.

DETAILED DESCRIPTION:
This study was planned as a single-dose, open label phase (Phase A) followed by a multiple-dose, double-blind, randomised, placebo-controlled, two-way crossover phase (Phase B) study in patients taking phenytoin. Phase B consisted of two 14-day treatment periods separated by a washout period of 10 to 15 days. Subjects continued their usual phenytoin scheme and received a single dose of ESL 1200 mg (Phase A) and either ESL (600 mg from Day 1 to 7 and 1200 mg from Day 8 to 14) or matching placebo once-daily for 14 days in each period.

The study was prematurely terminated due to impossibility of recruiting the planned number of patients. Only 4 patients were admitted and this was considered a too small sample size to allow a reliable assessment of the potential interaction between ESL and phenytoin. Therefore, no pharmacokinetic evaluation was performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 65 years, inclusive.
* Subjects who were on an established regimen of phenytoin monotherapy, which had been stable for at least 3 months.
* Subjects who had clinical laboratory tests acceptable to the Investigator.
* Subjects who were negative for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody (Ab) and human immunodeficiency viruses (HIV-1 and HIV-2) Ab tests at screening.
* Subjects who were negative for alcohol and drugs of abuse at screening.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to gave written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier or intrauterine device.
* (If female) She had a negative pregnancy test at screening.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of any disease that may interfere with the pharmacokinetics or pharmacodynamics of the Investigational Products, or may affect its safety.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse in the last 2 years.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had one of the following findings on the electrocardiogram (ECG): sinus bradycardia, sinoatrial block, atrioventricular block of any degree.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used any drugs (other than phenytoin) that may affect the pharmacokinetic profile of the investigational products within 2 weeks of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within 3 months of their first admission to this study.
* Subjects who had previously received ESL.
* Subjects who had donated and/or received any blood or blood products within the previous 3 months prior to screening.
* Subjects who were vegetarians, vegans and/or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to gave written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an approved effective contraceptive method.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2002-11; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events reported | 3 weeks
  Number of the adverse events reported

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Department, Hospital of Santa Maria, Lisbon, Lisbon District, Portugal